CLINICAL TRIAL: NCT07352865
Title: An Embedded Adaptive Randomized Controlled Trial of Corticosteroid Therapy for Severe Chlamydia Psittaci Community-Acquired Pneumonia in Adults
Brief Title: Adaptive RCT of Corticosteroids for Severe Chlamydia Psittaci Pneumonia in Adults
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Qingyuan Zhan (Other)
Responsible Party: Sponsor-Investigator, Qingyuan Zhan, Director, China-Japan Friendship Hospital
Organization: China-Japan Friendship Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025-I2M-C&T-B-090D
Record Dates: First submitted 2026-01-13; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Psittacosis
Keywords: Psittacosis; community-acquired pneumonia; adaptive randomised controled trial; corticosteroids
MeSH Terms: conditions — Psittacosis; Community-Acquired Pneumonia | interventions — Sodium Chloride; Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of Care (Placebo Comparator): Control group
  Interventions: Drug: Saline (0.9%, sterile, for infusion)
- Low dose steroids (Experimental): treated with low dose corticosteroids
  Interventions: Drug: low dose Methylprednisolone
- Moderate dose steroids (Experimental): treated with moderate dose corticosteroids
  Interventions: Drug: Moderate dose Methylprednisolone

INTERVENTIONS:
Drug: Saline (0.9%, sterile, for infusion) — Sailine as control
  Arms: Standard of Care
Drug: low dose Methylprednisolone — Methylprednisolone 0.5mg/kg ivgtt qd
  Arms: Low dose steroids
Drug: Moderate dose Methylprednisolone — Methylprednisolone 1.0mg/kg ivgtt qd
  Arms: Moderate dose steroids

SUMMARY:
Severe community-acquired pneumonia caused by psittacosis is a form of atypical-pathogen community-acquired pneumonia that often requires critical care management. It can occur in immunocompetent adults, has an abrupt onset and rapid progression, and may quickly deteriorate to profound hypoxemia, acute respiratory distress syndrome, and multiple organ dysfunction, frequently necessitating ICU admission. In a multicenter cohort from 19 tertiary hospitals in China with metagenomic next-generation sequencing (mNGS)-confirmed severe CAP complicated by acute hypoxemic respiratory failure, approximately 44% of patients required invasive mechanical ventilation and ICU mortality was 8.9%, indicating a substantial risk of death and severe morbidity among critically ill patients. The World Health Organization (WHO) reported an increase in cases across several European countries from 2023 to early 2024, with five deaths, suggesting that the disease burden and public health significance of psittacosis may have been underestimated for a prolonged period.

At present, the cornerstone of psittacosis pneumonia management is early recognition and timely pathogen-directed antibiotic therapy (tetracyclines, particularly doxycycline, as first-line treatment), together with well-established organ-support strategies. Optimizing comprehensive management beyond early standard supportive care and guideline-concordant antimicrobial therapy (including targeted antibiotics and organ support) to further reduce mortality in severe psittacosis pneumonia is therefore of major clinical importance for improving outcomes in critically ill patients and alleviating the burden on families and society. Accordingly, we plan to conduct an adaptive, randomized, open-label, controlled trial to evaluate the efficacy and safety of adjunctive corticosteroid regimens at different doses, in addition to early standard supportive care, for reducing mortality in patients with severe psittacosis pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Admission to the Intensive Care Unit (ICU).
* Meeting the diagnostic criteria for community-acquired pneumonia (CAP).
* Meeting at least one of the major diagnostic criteria for severe pneumonia:

  (i) Requirement for endotracheal intubation and mechanical ventilation;

(ii) Septic shock requiring vasopressor therapy after adequate fluid resuscitation.

-Or simultaneously fulfilling three of the minor criteria:

(i) Respiratory rate ≥ 30 breaths/min;

(ii) PaO₂/FiO₂ ≤ 250 mmHg;

(iii) Multilobar infiltrates;

(iv) Altered mental status and/or disorientation;

(v) Blood urea nitrogen ≥ 20 mg/dL (7.12 mmol/L);

(vi) Leukopenia (white blood cell count < 4 × 10⁹/L);

(vii) Thrombocytopenia (platelet count < 100 × 10⁹/L);

(viii) Hypothermia (core temperature < 36 °C);

(ix) Hypotension (systolic blood pressure < 90 mmHg) requiring aggressive fluid resuscitation.

* Confirmed Chlamydia psittaci etiology (psittacosis): at least one positive nucleic acid test (PCR/RT-PCR) or next-generation sequencing (NGS) result for Chlamydia psittaci in respiratory specimens (respiratory secretions, throat swabs, or bronchoalveolar lavage fluid).
* Severe community-acquired pneumonia (SCAP) patients admitted to the emergency department/ward/ICU due to respiratory failure within < 72 hours.
* Signed informed consent.

Exclusion Criteria:

* Patients receiving vasopressor therapy for septic shock at the time of enrollment.
* Terminally ill patients (expected survival <30 days, e.g., advanced malignancy).
* Clinical history suggesting overt aspiration.
* Documented active gastrointestinal bleeding.
* Presence of cystic fibrosis, obstructive pneumonia, active influenza, pulmonary tuberculosis, or fungal infection.
* Active viral hepatitis or active herpesvirus infection.
* Bone marrow suppression or HIV infection.
* Refusal of mechanical ventilation and endotracheal intubation.
* Uncontrolled hyperglycemia (diabetic ketoacidosis with blood ketones >3 mmol/L, or hyperosmolar hyperglycemic state with blood glucose >33.3 mmol/L and elevated osmolality).
* Known allergy to corticosteroids.
* Patients requiring anti-inflammatory corticosteroids or replacement hydrocortisone for any reason, or those already receiving prednisone >15 mg/day (or equivalent dose of another corticosteroid).
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
28-day all cause mortality | 28 days from inclusion

IPD SHARING:
Plan to Share IPD: Undecided